CLINICAL TRIAL: NCT05862155
Title: Prediction of Vesicouterine Adhesions by the Real-time Dynamic Transvaginal Sonographic Sliding Sign Technique: a Validation Study
Brief Title: Prediction of Vesicouterine Adhesions by Transvaginal Sonographic Sliding Sign Technique: a Validation Study
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, J.A.F. Huirne, Prof. Dr. J.A.F. Huirne, Amsterdam UMC, location VUmc
Other Study IDs: Sliding Bladder
Record Dates: First submitted 2023-05-05; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Adhesions Pelvic; Adhesion; Uterus; Adhesion; Bladder
Keywords: adhesion; vesicouterine; bladder; uterus; real-time dynamic; transvaginal sonography; sliding sign; ultrasound
MeSH Terms: conditions — Gynatresia; Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the predictive value of the real-time dynamic TVS sliding sign for vesicouterine pouch adhesions in women and to test the inter- and intraobserver agreement of this new technique.

DETAILED DESCRIPTION:
The investigators will conduct a prospective observational double-blind cohort study of patients who will have laparoscopic abdominopelvic surgery between January 2020 and December 2022 in the Amsterdam UMC. All women will be examined by TVE ultrasounds prior to surgery. The investigators will evaluate the predictive value of the real-time dynamic TVS sliding sign for vesicouterine pouch adhesions in women and test the inter- and intraobserver agreement of this technique.

All real-time dynamic transvaginal ultrasounds will be performed as followed: By mild pressure with the vaginal probe in the anterior vagina and palpation on the fundus with the free hand, the uterus will be pushed away from the bladder. The sliding-sign will be considered to be positive when the anterior wall glided freely in relation tot the bladder, one against the other. The sliding-sign was negative when the bladder is fixated tot the uterus for more than 1 cm from the vesico-vaginal fold. Or when the distance between the vesico-vaginal fold and the vesico-uterine fold is > 1 cm.

Two experienced gynaecologists and one resident in gynecology and obstetrics will evaluate the ultrasounds on the presence of the sliding sign independent from each other and without any knowledge of the individual patient and laparoscopic footage. All ultrasounds will be coded, so the assessors are blinded for the patients demographics and surgical history in order to interpret the sliding sign objectively.

The recorded laparoscopic videoclips will be evaluated by one of the researchers without any knowledge of the individual patient, surgical history and ultrasounds. Therefore the laparoscopic footage will be coded. To prevent bias the assessor will be blinded to the results of the ultrasound sliding sign assessments. Adhesions between uterus and bladder, abdominal fascia and omentum are scored according the classification of Tulandi. An adhesion score of 0 will be classified as no adhesions and an adhesion score of >16 as a 'frozen bladder'.

The obtained data will be analyzed to determine the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the sliding sign to predict the presence of absence of adhesions between the bladder and uterus. Fisher's exact test will be used to calculate the p-value for prediction of adhesions using the sliding sign technique. A P < 0.05 will be considered statistically significant. Interobserver variability will be assesed between two experienced gynecologists and between one experienced gynecologist and the resident. To assess the intraobserver variability one of the experienced gynecologists will reevaluated the same ultrasounds 2 months after the first ultrasound evaluation.

The investigators will try to obtain 100 inclusions based on previous studies who studied the role of the abdominal sonographic sliding sign in predicting intra-abdominal adhesions in pregnant women undergoing repeat cesarean section. All women have signed an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years old
* Laparoscopic abdominopelvic surgery with available video footage in Clinical Assistent
* Recorded real-time dynamic transvaginal ultrasound with the sliding sign technique
* Signed informed consent

Exclusion Criteria:

* Insufficient quality of the ultrasound
* Unclear laparoscopic videoclip to determine the presence of adhesions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing laparoscopic gynecological surgery at the Amsterdam UMC, location AMC who signed informed consent for the Status Studies, Niche Cohort or QUESTA study.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Transvaginal sonographic sliding sign | Preoperative
  Real-time dynamic transvaginal sonographic sliding sign (positive or negative sign)

SECONDARY OUTCOMES:
Adhesion score | Intraoperative recording of laparoscopic footage with postoperative assessment of the adhesion score based on this video within 2 years
  Adjusted classification of adhesions between uterus and bladder, abdominal fascia and omentum during laparoscopy. Total adhesion score of 0 = no adhesions. Total adhesion score of >16 = 'Frozen Bladder'.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Huirne, Prof. Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baron J, Tirosh D, Mastrolia SA, Ben-Haroush Y, Schwartz S, Kerner Y, Hershkovitz R. Sliding sign in third-trimester sonographic evaluation of intra-abdominal adhesions in women undergoing repeat Cesarean section: a novel technique. Ultrasound Obstet Gynecol. 2018 Nov;52(5):662-665. doi: 10.1002/uog.19057. PMID 29575202
- [Background] Hudelist G, Oberwinkler KH, Singer CF, Tuttlies F, Rauter G, Ritter O, Keckstein J. Combination of transvaginal sonography and clinical examination for preoperative diagnosis of pelvic endometriosis. Hum Reprod. 2009 May;24(5):1018-24. doi: 10.1093/humrep/dep013. Epub 2009 Feb 6. PMID 19202143
- [Background] Tulandi T, Lyell DJ. Classification of intra-abdominal adhesions after cesarean delivery. Gynecol Surg. 2013;10(1):25-9.
- [Derived] Min N, van Keizerswaard J, Visser RH, Burger NB, Rake JWT, Aarts JWM, Van den Bosch T, Leonardi M, Huirne JAF, de Leeuw RA. Prediction of vesicouterine adhesions by transvaginal sonographic sliding sign technique: validation study. Ultrasound Obstet Gynecol. 2025 Jan;65(1):114-121. doi: 10.1002/uog.29128. Epub 2024 Nov 25. PMID 39587459